CLINICAL TRIAL: NCT04933903
Title: BrUOG 397: NEO Rad (LOW): Neoadjuvant Low Dose Stereotactic Body Radiotherapy, Ipilimumab and Nivolumab for Patients With Resectable Stage IB - III Non-Small Cell Lung Cancer
Brief Title: BrUOG 397: NEO Rad (LOW): Neoadjuvant Low Dose Stereotactic Body Radiotherapy, Ipilimumab and Nivolumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 397
Record Dates: First submitted 2020-10-15; First posted 2021-06-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Protocol Therapy (Experimental): Ipilimumab: 1mg/kg IV day 1. Nivolumab: 3mg/kg IV days 1, 15, 29. SBRT delivered as 1-2 fractions to the gross primary tumor and nodal disease following day 1 infusion and completed by day 3 (7Gy x 1; 4Gy x 2).
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Radiation: SBRT

INTERVENTIONS:
Drug: Ipilimumab — 1mg/kg IV on day 1 (1 dose total)
Drug: Nivolumab — 3mg/kg (to a maximum of 240mg) IV on days 1, 15, 29 (+/- 3 days) (3 doses total)
Radiation: SBRT — 1 fraction or 2 fractions delivered to the gross primary tumor and nodal disease, following the first treatment with ipilimumab + nivolumab on days 1-3.

SUMMARY:
This single-arm phase 2 study will enroll patients with resectable and operable stage IB - III non-small cell lung cancer and treat them with pre-operative ipilimumab + nivolumab plus low-dose stereotactic body radiation therapy (SBRT) delivered concurrently. Only patients who proceed to surgery will be evaluable for the primary endpoint. The primary efficacy outcome measurement will be pathologic response (including Major Pathologic Response (MPR), and Complete Pathologic Response (CPR)). Secondary outcome measures include safety, and exploratory biomarkers of immune response in pre- and post-operative blood and tissue. A two-stage design will stop the study if fewer than 3 of the first 9 evaluable patients do not achieve MPR. An early stopping rule for safety will stop the study if more than 12 patients are enrolled to find the first 9 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed NSCLC
2. Age > 18
3. ECOG Performance Status 0-1.
4. Pulmonary function capacity capable of tolerating the proposed lung resection. FEV1 at least 2 L. If less than 2 L, the predicted postoperative forced expiratory volume in 1 second (FEV1) must be > 0.8 L or be > 35% of the predicted value. Postoperative predicted DLCO ≥ 35% is required.
5. Resectable stage IB-IIIB (T2-3N0, T1-T3N1-2) NSCLC (per the 8th Edition American Joint Committee on Cancer (AJCC) classification) who are candidates for surgery with intent of R0 resection. Invasive T3 disease (eg, phrenic nerve, pericardium, chest wall other than Pancoast superior sulcus) may be included if the surgeon and study team deem it to be resectable.
6. N2 nodes must be discrete (ie, not invading surrounding structures). If patients have N2 disease, as suspected by CT or PET, histologic proof of N2 status is recommended.
7. Patients must be evaluated by a Thoracic Surgeon prior to registration. Operability is defined as having adequate pulmonary, cardiac, renal, nutritional, musculoskeletal, neurologic, and cognitive capacity to undergo major pulmonary resection with acceptable morbidity and mortality. Absence of major associated comorbidities that increase the surgery risk to an unacceptable level.
8. No prior history of thoracic radiation.
9. Adequate Organ and marrow function as defined below

   * leukocytes ≥2,000/mcL,
   * absolute neutrophil count ≥1,000/mcL,
   * platelets ≥100,000/mcL,
   * Hemoglobin >8.0 g/dL
   * Total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
   * creatinine within normal institutional limits OR creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
10. Patients are capable of giving informed consent and/or have an acceptable surrogate capable of giving consent on the subject's behalf.
11. Nonpregnant and non-nursing. The effect of ipilimumab and nivolumab on the fetus is unknown.
12. Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses >1 year.
13. Evidence of postmenopausal status or negative urinary or serum pregnancy test for female premenopausal patients. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
14. Women <50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
15. Women ≥50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
17. Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.

Exclusion Criteria:

1. Pathologically confirmed NSCLC *
2. Age > 18 *
3. ECOG Performance Status 0-1.
4. Pulmonary function capacity capable of tolerating the proposed lung resection. FEV1 at least 2 L. If less than 2 L, the predicted postoperative forced expiratory volume in 1 second (FEV1) must be > 0.8 L or be > 35% of the predicted value. Postoperative predicted DLCO ≥ 35% is required.
5. Resectable stage IB-IIIB (T2-3N0, T1-T3N1-2) NSCLC (per the 8th Edition American Joint Committee on Cancer (AJCC) classification) who are candidates for surgery with intent of R0 resection. Invasive T3 disease (eg, phrenic nerve, pericardium, chest wall other than Pancoast superior sulcus) may be included if the surgeon and study team deem it to be resectable.
6. N2 nodes must be discrete (ie, not invading surrounding structures). If patients have N2 disease, as suspected by CT or PET, histologic proof of N2 status is recommended.
7. Patients must be evaluated by a Thoracic Surgeon prior to registration. Operability is defined as having adequate pulmonary, cardiac, renal, nutritional, musculoskeletal, neurologic, and cognitive capacity to undergo major pulmonary resection with acceptable morbidity and mortality. Absence of major associated comorbidities that increase the surgery risk to an unacceptable level. *
8. No prior history of thoracic radiation.
9. Adequate Organ and marrow function as defined below

   * leukocytes ≥2,000/mcL,
   * absolute neutrophil count ≥1,000/mcL,
   * platelets ≥100,000/mcL,
   * Hemoglobin >8.0 g/dL
   * Total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
   * creatinine within normal institutional limits OR creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
10. Patients are capable of giving informed consent and/or have an acceptable surrogate capable of giving consent on the subject's behalf.
11. Nonpregnant and non-nursing. The effect of ipilimumab and nivolumab on the fetus is unknown.
12. Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses >1 year.
13. Evidence of postmenopausal status or negative urinary or serum pregnancy test for female premenopausal patients. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
14. Women <50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
15. Women ≥50 years of age would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
17. Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with a Pathologic Response | From beginning of study treatment to approximately day 49-63 on study.
  Assess Pathologic Response (major pathologic response and complete pathologic response) following neoadjuvant low dose SBRT, Ipilimumab and Nivolumab.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Beginning of study treatment through 90 days post study treatment completion.
  Assess safety and operative morbidity following neoadjuvant low dose SBRT, Ipilimumab and Nivolumab and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Azzoli, MD, Principal Investigator — Brown University; Thomas A DiPetrillo, MD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States